CLINICAL TRIAL: NCT04437498
Title: Non-Invasive Vagal Nerve Stimulation in Veterans With Mild Traumatic Brain Injury (mTBI)
Brief Title: Vagal Nerve Stimulation in mTBI
Acronym: VNS mTBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N3418-I; I01RX003418 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: PTSD; mTBI
Keywords: vagus nerve; stress disorders, posttraumatic; traumatic brain injury; memory; hippocampus; emission tomography
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Veterans are randomized to double blind treatment with active non-invasive Vagal Nerve Stimulation (nVNS) or a sham control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: code for active and sham devices kept by non study personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- nVNS (Experimental): non invasive vagal nerve stimulation
  Interventions: Device: nVNS
- sham (Sham Comparator): sham stimulation
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: sham stimulation — non invasive vagal nerve stimulation
  Arms: sham
Device: nVNS — active vns stimulation
  Arms: nVNS

SUMMARY:
Mild traumatic brain injury (mTBI) and posttraumatic stress disorder (PTSD) are important conditions for the Veterans Administration (VA) that frequently occur together in combat Veterans from the conflicts in Afghanistan and Iraq. In many Veterans these become chronic, raising the risk the burden of neurotrauma can worsen over time. This study will examine a new intervention called non-invasive Vagal Nerve Stimulation (nVNS) and its effects on memory and symptoms of PTSD and mTBI as well as brain and physiology in Veterans with mTBI and PTSD.

DETAILED DESCRIPTION:
This projects will assess the effects of non-invasive Vagal Nerve Stimulation (nVNS) on neurobiology and cognition in combat Veterans with mild Traumatic Brain Injury (mTBI) and co-morbid posttraumatic stress disorder (PTSD) during the performance of stressful tasks (traumatic scripts, mental arithmetic) and verbal declarative memory tasks using measurement of memory performance, peripheral inflammatory markers in blood (IL6) and cardiovascular responses using wearable gated sensing devices and electro- and seismocardiography, as well as brain response (anterior cingulate, hippocampus) measured with High Resolution Positron Emission Tomography (HR-PET) and radiolabelled water (15O[H2O]). The investigators hypothesize that nVNS but not sham control will result in enhanced memory, and hippocampal activation with memory encoding, and reduced cardiovascular, sympathetic, and inflammatory responses to stress. The investigators will also assess the effects of nVNS and sham on memory retention when applied to the encoding phase of a declarative memory learning task repeated daily over a four day period and on ratings of PTSD and pain in Veterans with mTBI and co-morbid PTSD and repeat assessments after three months of twice daily treatments.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with mTBI and PTSD

Exclusion Criteria:

* amnesia for the inciting event lasted longer than 24 hours
* Glasgow Coma Scale Score after 30 minutes was less than 13
* loss of consciousness more than 30 minutes
* positive pregnancy test
* meningitis or other neurological disorder other than mTBI
* alcohol or substance abuse use disorder based on the SCID within the past 12 months
* current or lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, anorexia nervosa or bulimia, based on the SCID
* active suicidal ideation based on criteria outlined below
* a history of serious medical or neurological illness, such as cardiovascular, gastrointestinal, hepatic, renal, neurologic or other systemic illness
* active neuroleptic, opiate, or benzodiazepine treatment
* structural abnormality on brain MRI or CT

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
CAPS | three months
  The Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale (CAPS) is a measure of PTSD symptoms with a range of 0-80 and higher score indicating more severe PTSD symptoms. We will compare change from baseline to post treatment with active vagal nerve stimulation (VNS) or sham stimulation twice daily.
insula | 10 minutes
  Blood flow in the insula is measured with positron emission tomography (PET) and radiolabelled water during the performance of stress tasks. We compare blood flow in the insula to whole brain blood flow ratio during stress tasks (listening to personalized traumatic scripts) versus control tasks in the VNS versus sham groups with hypothesis of blocked insula blood flow with VNS
HVLT-R % retention | baseline versus three months
  The Hopkins Verbal Learning Test-Revised (HVLT-R) is a test of declarative memory learning that involves the learning of 12 nouns, four from each of three semantic categories, learned over three learning trials, followed 20 minutes later by a delayed free recall trial and recognition trial composed of 24 words with 12 false positives. The percent (%) retention is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3. HLVT-R % retention has a range of 0-100 with 100 being best and 0 worst performance. Baseline and three months post treatment paired with sham or active stimulation are compared.
Change in IL6 Concentration in Blood with Stress | Baseline to 120 minutes after stress
  Interleukin-6 (IL6) response to stress paired with active or sham stimulation. IL6 is an inflammatory biomarker measured in blood. We compare IL6 response to stress in VNS versus sham treated groups.
hippocampal activation | 10 minutes
  Blood flow in the hippocampus is measured with positron emission tomography (PET) and radiolabelled water during the performance of declarative memory tasks. We compare blood flow in the hippocampus to whole brain blood flow ratio during memory tasks versus control tasks in the VNS versus sham groups with hypothesis of increased hippocampal blood flow with VNS

SECONDARY OUTCOMES:
PPG amplitude | Change from baseline to 5 seconds after the termination of stimulation paired with stress
  Photoplethysmography (PPG) amplitude is a measure of peripheral vasoconstriction which is a marker of sympathetic response to stress with active or sham. PPG amplitude is the diameter of the blood vessel in the finger, we measure change from baseline to post active vagal nerve stimulation versus sham stimulation with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Doug J Bremner, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: three months after study end
Access Criteria: de identified data for three years